CLINICAL TRIAL: NCT04234074
Title: Improved Discrimination Of Central And Obstructive Apnoeas In Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH/13/023
Record Dates: First submitted 2015-12-04; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Central And Obstructive Apnoeas In Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Breathing test or sleep study (Other): infants undertaking cardiorespiratory polysomnography
  Interventions: Device: Volusense paediatric monitoring device

INTERVENTIONS:
Device: Volusense paediatric monitoring device — Comparison of Volusense paediatric monitoring device to full cardiorespiratory polysomnography.
  Other Names: Volusense

SUMMARY:
Referral of infants to the respiratory sleep disorders breathing team with apnoeas [pauses in their breathing] and apparent life-threatening episodes are frequent. While the majority of such episodes do not have a significant underlying problem a potentially life threatening condition accounts for a significant proportion of cases.

In order to fully assess an infant, a full-scale overnight polysomnography study would be required. Unfortunately due to the complexity of such studies and because the equipment is generally fully booked for many weeks ahead it is extremely difficult to arrange timely assessment. Hence, currently, we are largely reliant on simple screening with pulse oximetry (measuring oxygen levels in the blood with a simple probe). This is able to identify potentially significant problems, but it is does not help to determine whether this is because the baby simply stops breathing for a period due to disturbance of its control of breathing, or whether it is experiencing obstructive episodes, for which there are a number of causes. This new equipment to be assessed would potentially provide a simple, robust means of undertaking definitive studies simply and effectively on the medical wards with assessment of chest and abdominal wall movement being linked to pulse oximetry.

This is likely to provide a substantial and significant improvement on our current practice. The benefits will be that, for those with no significant underlying problems, we will be able to provide much greater reassurance for the parents, which is clearly very valuable, while in those with a problem we will be able to distinguish those with central or obstructive apnoea with a degree of certainty that will greatly streamline further assessments and treatment.

ELIGIBILITY:
Inclusion Criteria:

•Infants between 36 weeks post conception and one year old referred to the respiratory and sleep team for central or obstructive apnoea or apparent life threatening events.

Exclusion Criteria:

•Chest wall deformity on injury that precludes the use of the Volusense paediatric device.

Ages: 36 Weeks to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Whether comparable to gold standard - cardiorespiratory polysomnogram | 74 months
  To measure the number of central apnoeas, obstructive apnoeas and hyponeas recorded and measured through the night. The apnoea/hyponea index will then be calculated

SECONDARY OUTCOMES:
To find if Volusense detects central and obstructive apnoea | 74 months
  To measure the number of central apnoeas, obstructive apnoeas and hyponeas recorded and measured through the night. The apnoea/hyponea index will then be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Kelechi Ugonna, Principal Investigator — Investigator
Locations (1):
- Sheffield Children's NHS Foundation Trust, Sheffield, Sheffield (South Yorkshire District), United Kingdom